CLINICAL TRIAL: NCT03158051
Title: The MyHEART Study: A Young Adult Hypertension Self-Management Randomized Controlled Trial
Brief Title: Young Adult Hypertension Self-Management Clinical Trial
Acronym: MyHEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-0372; R01HL132148 (NIH); A534225 (Other: UW Madison); SMPH\MEDICINE\CARDIOLOGY (Other: UW Madison)
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Hypertension; Blood Pressure; Lifestyle Risk Reduction
Keywords: Hypertension; Young Adult; Self-Management; Health coach
MeSH Terms: conditions — Hypertension; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Telephone health coaching, home blood pressure monitoring, individualized goal setting, and tailored educational materials
  Interventions: Behavioral: Home Blood Pressure Monitoring; Behavioral: Telephone Health Coaching
- Usual clinical care (No Intervention): Usual care arm participants will receive routine hypertension clinical care per their primary care provider.

INTERVENTIONS:
Behavioral: Home Blood Pressure Monitoring — Intervention arm participants will receive a home blood pressure monitor, home blood pressure log, and training on accurate home monitoring. They will be asked to share their home blood pressure readings during health coach telephone calls.
  Arms: Intervention
Behavioral: Telephone Health Coaching — Intervention arm participants will receive a health coach phone call every 2 weeks for 6 months, for a total of 12 calls. During each call, the health coach will review and discuss home blood pressures and address barriers and concerns to hypertension management. During each telephone call, the coach will guide the participant on selecting health behavior goals. Intervention arm participants will also receive handouts about hypertension management during the study visits and after health coach calls.
  Arms: Intervention

SUMMARY:
This is a 5-year randomized controlled trial in two large healthcare systems (Madison and Milwaukee, WI) to evaluate MyHEART's (My Hypertension Education And Reaching Target) impact on blood pressure among 310 geographically and racially/ethnically diverse young adults.

DETAILED DESCRIPTION:
Aim 1. To evaluate the effect of MyHEART (home blood pressure monitor distribution and heath coaching) on clinical outcomes, the change in systolic and diastolic blood pressure (primary) and hypertension control (secondary) after 6 and 12 months, compared to usual clinical care.

Aim 2. To evaluate the effect of MyHEART on hypertension self-management behavior (behavioral outcomes) at 6 and 12 months, compared to usual clinical care.

Aim 3. To examine whether MyHEART's effects on self-management behavior are mediated through variables of perceived competence, autonomy, motivation, and activation (mediation outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable of giving written informed consent
* Willing to comply with all study procedures and be available for the duration of the study
* Males and females ages 18-39 years old at the start of the study (inclusive)
* A minimum of two hypertension ICD-10 coded visits with a provider (physician [MD, DO], physician assistant, nurse practitioner) on different dates in the last 24 months, with at least one code in the past 18 months
* Medically homed at an IRB approved healthcare system

Exclusion Criteria:

* History of medically determined Congestive Heart Failure
* Unable to provide informed consent (i.e., activated healthcare power of attorney)
* Unable or unwilling to travel to local clinic for research visits
* Currently residing in a skilled nursing facility
* Diagnosed with sickle cell anemia or cystic fibrosis
* Diagnosed with stroke, myocardial infarction, and/or coronary artery revascularization in the past 2 years
* Syncope while exercising or doing strenuous activity within past 12 months
* Currently prescribed warfarin, novel oral anticoagulant, or insulin
* Planned organ transplant or prior transplant in the past 5 years
* Chemotherapy or radiation therapy within 6 the past months
* Severely impaired hearing, vision, or speech, as determined by study staff responsible for enrollment
* Current participation or planning to participate in another clinical trial in the next 12 months
* Pregnant or planning to become pregnant in the next 12 months
* Planning to leave the geographic area in the next 6 months
* Health condition that will limit both increasing physical activity and changing diet
* Illegal drug use (other than marijuana) in the past 30 days
* Unable to read or communicate in English
* Currently on dialysis or seeing a Nephrologist
* Unaware or denies history of high blood pressure or hypertension
* Between-arm blood pressure difference >20 mmHg
* White Coat Hypertension (24-hour ambulatory monitoring)
* Inability to comply with or complete the protocol or other reasons at the discretion of the principal and site investigators
* Prisoners

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 316 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara Hoppe, DO, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin School of Medicine & Public Health, Madison, Wisconsin
  - Aurora Health Care, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson HM, Sullivan-Vedder L, Kim K, McBride PE, Smith MA, LaMantia JN, Fink JT, Knutson Sinaise MR, Zeller LM, Lauver DR. Rationale and study design of the MyHEART study: A young adult hypertension self-management randomized controlled trial. Contemp Clin Trials. 2019 Mar;78:88-100. doi: 10.1016/j.cct.2019.01.010. Epub 2019 Jan 21. PMID 30677485
- [Derived] Hoppe KK, Smith M, Birstler J, Kim K, Sullivan-Vedder L, LaMantia JN, Knutson Sinaise MR, Swenson M, Fink J, Haggart R, McBride P, Lauver DR, Johnson HM. Effect of a Telephone Health Coaching Intervention on Hypertension Control in Young Adults: The MyHEART Randomized Clinical Trial. JAMA Netw Open. 2023 Feb 1;6(2):e2255618. doi: 10.1001/jamanetworkopen.2022.55618. PMID 36735261

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Usual Clinical Care
Started | 157 | 159
Visit 3 | 100 | 104
Visit 4 | 100 | 104
Visit 5 | 86 | 90
Visit 6 | 86 | 89
Completed | 86 | 89
Not Completed | 71 | 70
Not completed — Lost to Follow-up | 41 | 47
Not completed — Physician Decision | 6 | 7
Not completed — Withdrawal by Subject | 24 | 15
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Clinical Care | Total
Number analyzed (Participants) | 157 | 159 | 316
Age, Continuous [Median (Full Range); unit: years] | 33.8 [18.0 to 39.0] | 33.7 [19.0 to 39.0] | 33.8 [18.0 to 39.0]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 71 | 74 | 145
  Male | 81 | 85 | 166
  Unknown | 5 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 37 | 35 | 72
  Other | 13 | 9 | 22
  White | 107 | 115 | 222
Region of Enrollment [Number; unit: participants]
  United States | 157 | 159 | 316
Alcohol Beverages per week [Median (Full Range); unit: servings of alcohol per week] | 5.3 [0.0 to 25.0] | 5.1 [0.0 to 32.0] | 5.2 [0.0 to 32.0]
Ambulatory Diastolic Blood Pressure (BP) [Median (Full Range); unit: mmHg] | 86.5 [68.0 to 110.0] | 87.0 [72.0 to 120.0] | 86.7 [68.0 to 120.0]
Ambulatory Systolic BP [Median (Full Range); unit: mmHg] | 132.6 [108.0 to 172.0] | 133.0 [112.0 to 183.0] | 132.8 [108.0 to 183.0]
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 34.5 [19.8 to 63.1] | 34.5 [19.3 to 57.8] | 34.5 [19.3 to 63.1]
Number of Children at Home [Median (Full Range); unit: children] | 1.1 [0.0 to 6.0] | 1.0 [0.0 to 6.0] | 1.0 [0.0 to 6.0]
Office Diastolic BP [Median (Full Range); unit: mmHg] | 90.8 [68.7 to 131.7] | 91.8 [66.0 to 136.3] | 91.3 [66.0 to 136.3]
Office Systolic BP [Median (Full Range); unit: mmHg] | 138.3 [106.0 to 185.3] | 138.0 [109.7 to 192.0] | 138.1 [106.0 to 192.0]
Waist Circumference [Median (Full Range); unit: centimeters] | 109.5 [65.0 to 178.0] | 109.4 [66.0 to 153.0] | 109.4 [65.0 to 178.0]
Weight [Median (Full Range); unit: kilograms] | 103.1 [53.0 to 206.0] | 103.3 [45.0 to 200.0] | 103.2 [45.0 to 206.0]
Cigarette Tobacco Status [Count of Participants; unit: Participants]
  Currently Smoke Cigarettes | 21 | 19 | 40
  Have Never Smoked Cigarettes | 97 | 115 | 212
  Used to Smoke Cigarettes | 34 | 25 | 59
  Unknown | 5 | 0 | 5
Godin-Shephard Physical Activity [Count of Participants; unit: Participants]
  Active | 68 | 81 | 149
  Insufficiently Active | 84 | 78 | 162
  Unknown | 5 | 0 | 5
Highest Level of Education [Count of Participants; unit: Participants]
  I have not finished High School | 7 | 8 | 15
  I have completed High School | 22 | 20 | 42
  I have not finished College or Vocational School | 28 | 24 | 52
  I have finished College or Vocational School | 63 | 74 | 137
  Some / Completed Graduate of Professional School | 32 | 33 | 65
  Unknown | 5 | 0 | 5
Marital Status [Count of Participants; unit: Participants]
  Single | 50 | 54 | 104
  Married / Partnered | 99 | 101 | 200
  Divorced / Widower | 3 | 4 | 7
  Unknown | 5 | 0 | 5
Number of Antihypertensive Medications [Count of Participants; unit: Participants]
  0 | 84 | 78 | 162
  1 | 46 | 51 | 97
  2 | 22 | 21 | 43
  3 | 3 | 8 | 11
  greater than or equal to 4 | 2 | 1 | 3
Self-Perceived Health Status [Count of Participants; unit: Participants]
  Excellent | 3 | 4 | 7
  Very Good or Good | 70 | 83 | 153
  Fair | 61 | 50 | 111
  Poor or No Response | 18 | 21 | 39
  Unknown | 5 | 1 | 6
Comorbidities [Count of Participants; unit: Participants]
  Anxiety and / or Depression | 82 | 78 | 160
  Chronic Kidney Disease | 1 | 2 | 3
  Diabetes | 9 | 9 | 18
  Dyslipidemia | 41 | 32 | 73
  Other Chronic Comorbidity | 62 | 59 | 121
Risk Factors [Count of Participants; unit: Participants]
  E-Cigarette / Vaping Use in the past 6 months | 13 | 13 | 26
  Ever Been on Medicaid | 34 | 33 | 67
  Family History of Heart Disease or Stroke | 52 | 61 | 113
  Financial Status: Inadequate Income | 126 | 122 | 248

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Systolic Ambulatory Blood Pressure (mmHg)
Description: 24-hour Systolic Ambulatory Blood Pressure measured at baseline, 6 months, and 12 months.
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Median (Standard Deviation); unit: mmHg
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
mmHg
  baseline | 132.59 (11.36) | 133.01 (12.67)
  6 month: number analyzed (Participants) | 100 | 102
  6 month | 128.14 (11.36) | 130.69 (13.99)
  12 month: number analyzed (Participants) | 85 | 88
  12 month | 128.54 (11.95) | 129.47 (14.71)

2. Primary Outcome: 24-hour Diastolic Ambulatory Blood Pressure (mmHg)
Description: 24-hour Diastolic Ambulatory Blood Pressure measured at baseline, 6 months, and 12 months.
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
mmHg
  baseline | 86.45 (7.76) | 87.04 (8.16)
  6 months: number analyzed (Participants) | 100 | 102
  6 months | 84.61 (8.24) | 85.89 (9.19)
  12 months: number analyzed (Participants) | 85 | 88
  12 months | 85.34 (9.32) | 85.52 (9.43)

3. Primary Outcome: Clinic Systolic Blood Pressure (mmHg)
Description: Systolic Blood Pressure measured at baseline, 6 months, and 12 months.
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Median (Standard Deviation); unit: mmHg
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
mmHg
  baseline | 138.30 (14.27) | 137.97 (14.33)
  6 month: number analyzed (Participants) | 100 | 104
  6 month | 130.84 (12.16) | 132.50 (15.83)
  12 month: number analyzed (Participants) | 86 | 90
  12 month | 131.16 (12.77) | 130.7 (15.22)

4. Primary Outcome: Clinic Diastolic Blood Pressure (mmHg)
Description: Clinic Diastolic Blood Pressure measured at baseline, 6 months, and 12 months.
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
mmHg
  baseline | 90.81 (11.42) | 91.77 (11.26)
  6 months: number analyzed (Participants) | 100 | 104
  6 months | 83.83 (9.36) | 86.70 (12.44)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 85.05 (10.56) | 85.15 (12.31)

5. Secondary Outcome: Number of Participants That Achieve Hypertension Control at 6 Months
Description: Hypertension Control: Percentage of participants that achieve hypertension control at 6 months. Hypertension control will be defined using ambulatory blood pressures as the gold standard (<130/80 mmHg); otherwise a clinic blood pressure of <140/90 mmHg will be used.
Time Frame: up to 6 months
Population: participants lost to follow up, withdrew, and/or removed from study per physician, 2 participants in the Usual clinical care arm did not wear their cuff long enough to get adequate readings for AMBP
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
Participants
  24-hour Ambulatory Blood Pressure: number analyzed (Participants) | 100 | 102
  24-hour Ambulatory Blood Pressure | 20 | 21
  Clinic Measured Blood Pressure: number analyzed (Participants) | 100 | 104
  Clinic Measured Blood Pressure | 60 | 60

6. Secondary Outcome: Sodium Intake as Assessed by the Automated Self-Administered 24-hour Dietary Assessment
Description: Mean daily sodium intake (milligrams/day) at baseline, 6 months, and 12 months as assessed by the computer administered Automated Self-Administered 24-hour Dietary Assessment
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: milligrams per day
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
milligrams per day
  baseline: number analyzed (Participants) | 149 | 155
  baseline | 3512.82 (1765.59) | 3672.81 (1812.82)
  6 months: number analyzed (Participants) | 99 | 104
  6 months | 3354.72 (1365.75) | 3968.20 (1725.17)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 3682.94 (1874.53) | 4213.67 (1972.37)

7. Secondary Outcome: Number of Combined Fruit and Vegetable Servings as Assessed by the Automated Self-Administered 24-hour Dietary Assessment
Description: Mean number of combined fruit and vegetable servings measured at baseline, 6 months, and 12 months as assessed by the computer administered Automated Self-Administered 24-hour Dietary Assessment, reported in cups equivalent.
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: cups per day
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
cups per day
  baseline: number analyzed (Participants) | 149 | 155
  baseline | 2.34 (2.02) | 2.50 (1.98)
  6 months: number analyzed (Participants) | 99 | 104
  6 months | 2.43 (1.75) | 2.57 (1.89)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 2.50 (1.92) | 2.55 (1.88)

8. Secondary Outcome: Ounces of Whole Grain as Assessed by the Automated Self-Administered 24-hour Dietary Assessment
Description: Ounces of whole grain measured at baseline, 6 months, and 12 months as assessed by the computer administered Automated Self-Administered 24-hour Dietary Assessment
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: ounces per day
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
ounces per day
  baseline: number analyzed (Participants) | 149 | 155
  baseline | 0.61 (1.05) | 0.85 (1.41)
  6 months: number analyzed (Participants) | 99 | 104
  6 months | 0.88 (1.49) | 1.12 (1.62)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 0.82 (1.25) | 1.14 (2.24)

9. Secondary Outcome: Saturated Fat as Assessed by the Automated Self-Administered 24-hour Dietary Assessment
Description: Saturated fat measured at baseline, 6 months, and 12 months as assessed by the computer administered Automated Self-Administered 24-hour Dietary Assessment, reported in percent kilocalories
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: percent kilocalories
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
percent kilocalories
  baseline: number analyzed (Participants) | 149 | 155
  baseline | 11.91 (4.19) | 12.54 (4.32)
  6 months: number analyzed (Participants) | 99 | 104
  6 months | 12.97 (4.62) | 13.12 (6.56)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 12.03 (4.72) | 13.46 (4.52)

10. Secondary Outcome: Physical Activity as Assessed by the Godin Physical Activity Questionnaire
Description: Mean weekly amounts of physical activity as assessed by the Godin Physical Activity Questionnaire. The Godin Physical Activity Questionnaire measures a person's strenuous, moderate, and light physical activity in a week. Scoring is calculated as follows (units are times per week that the participant engaged in any of the 3 classifications of activity longer than 15 minutes during their free time):
  * 9 x strenous units reported + 5 x moderate units reported + 3 x light units reported = score
  A minimum score of 0 indicates no activity, a score of less than 14 is interpreted as insufficiently active or sedentary, a score between 14 and 23 is interpreted to be moderately active, and a score of 24 and higher is interpreted to be active, a theoretical maximum does not exist.
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
score on a scale
  baseline: number analyzed (Participants) | 152 | 159
  baseline | 38.24 (31.51) | 37.24 (26.99)
  6 months: number analyzed (Participants) | 100 | 104
  6 months | 54.47 (61.99) | 40.69 (31.80)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 46.67 (46.10) | 39.22 (25.22)

11. Secondary Outcome: Home Blood Pressure Monitoring Frequency
Description: Self-report of home blood pressure monitoring frequency measured at baseline, 6 months, and 12 months.
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
Participants
  Baseline: number analyzed (Participants) | 152 | 159
  Baseline: Not on a regular basis | 109 | 118
  Baseline: At least once per month | 23 | 20
  Baseline: At least once a week | 13 | 17
  Baseline: At least once a day | 7 | 4
  6 months: number analyzed (Participants) | 100 | 104
  6 months: Not on a regular basis | 14 | 67
  6 months: At least once per month | 9 | 22
  6 months: At least once a week | 64 | 10
  6 months: At least once a day | 13 | 5
  12 months: number analyzed (Participants) | 86 | 90
  12 months: Not on a regular basis | 32 | 67
  12 months: At least once per month | 20 | 11
  12 months: At least once a week | 30 | 8
  12 months: At least once a day | 4 | 4

12. Secondary Outcome: Standing Weight (kg)
Description: Weight (kg) measured at baseline, 6 months, and 12 months.
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
kilograms
  baseline: number analyzed (Participants) | 151 | 159
  baseline | 102.86 (28.64) | 102.93 (27.30)
  6 months: number analyzed (Participants) | 100 | 104
  6 months | 98.54 (26.19) | 103.80 (25.34)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 97.91 (26.07) | 103.45 (25.49)

13. Secondary Outcome: Perceived Competence as Assessed by the Perceived Competence Scale for Diet
Description: Perceived competence measured at baseline, 6 months, and 12 months as assessed by the Perceived Competence Scale (self-administration). This is a 4-item survey scored on a 7 point likert scale from 1 (not at all true) to 7 (very true). Mean score from 1-7 will be reported with higher scores indicating increased perceived competence.
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
score on a scale
  Baseline: number analyzed (Participants) | 152 | 159
  Baseline | 4.54 (1.34) | 4.56 (1.30)
  6 months: number analyzed (Participants) | 100 | 104
  6 months | 5.04 (1.24) | 4.63 (1.43)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 4.71 (1.25) | 4.70 (1.30)

14. Secondary Outcome: Perceived Competence as Assessed by the Perceived Competence Scale for Exercise
Description: as for outcome 13
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
score on a scale
  Baseline: number analyzed (Participants) | 152 | 159
  Baseline | 4.83 (1.45) | 5.03 (1.46)
  6 months: number analyzed (Participants) | 100 | 104
  6 months | 5.28 (1.37) | 5.01 (1.54)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 4.98 (1.47) | 4.89 (1.49)

15. Secondary Outcome: Perceived Autonomy as Assessed by the Health Care Climate Questionnaire for Diet
Description: Perceived autonomy measured at baseline, 6 months, and 12 months as assessed by the Health Care Climate Questionnaire (self-administration). This is a 6-item survey scored on a 7 point likert scale from 1 (not at all true) to 7 (very true). Mean between 1-7 will be reported with higher scores indicative of increased perceived autonomy.
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
score on a scale
  baseline: number analyzed (Participants) | 152 | 159
  baseline | 4.63 (1.60) | 4.93 (1.58)
  6 months: number analyzed (Participants) | 100 | 104
  6 months | 5.35 (1.41) | 5.17 (1.48)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 5.06 (1.52) | 5.22 (1.40)

16. Secondary Outcome: Perceived Autonomy as Assessed by the Health Care Climate Questionnaire for Exercise
Description: as for outcome 15
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
score on a scale
  baseline: number analyzed (Participants) | 152 | 159
  baseline | 4.72 (1.65) | 5.00 (1.53)
  6 months: number analyzed (Participants) | 100 | 104
  6 months | 5.31 (1.38) | 5.17 (1.50)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 5.11 (1.57) | 5.31 (1.40)

17. Secondary Outcome: Autonomous Motivation as Assessed by the Treatment Self-Regulation Questionnaire for Diet
Description: Autonomous motivation measured at baseline, 6 months, and 12 months as assessed by the Treatment Self-Regulation Questionnaire (self-administration). This is a 15-item survey scored on a 7 point likert scale from 1 (not at all true) to 7 (very true). Mean score between 1 and 7 will be reported with higher scores indicative of increased autonomous motivation.
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
score on a scale
  baseline: number analyzed (Participants) | 152 | 159
  baseline | 5.80 (1.02) | 5.80 (1.06)
  6 months: number analyzed (Participants) | 100 | 104
  6 months | 5.86 (1.02) | 5.76 (1.02)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 5.78 (1.02) | 5.85 (0.95)

18. Secondary Outcome: Autonomous Motivation as Assessed by the Treatment Self-Regulation Questionnaire for Exercise
Description: as for outcome 17
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
score on a scale
  baseline: number analyzed (Participants) | 152 | 159
  baseline | 5.81 (1.04) | 5.81 (1.07)
  6 months: number analyzed (Participants) | 100 | 104
  6 months | 5.94 (1.00) | 5.74 (1.03)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 5.79 (1.06) | 5.83 (1.04)

19. Secondary Outcome: Controlled Motivation as Assessed by the Treatment Self-Regulation Questionnaire for Diet
Description: Controlled motivation measured at baseline, 6 months, and 12 months as assessed by the Treatment Self-Regulation Questionnaire (self-administration). This is a 15-item survey scored on a 7 point likert scale from 1 (not at all true) to 7 (very true). Mean score between 1 and 7 will be reported with higher scores indicative of increased controlled motivation.
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
score on a scale
  baseline | 3.19 (1.25) | 3.04 (1.23)
  6 months: number analyzed (Participants) | 100 | 104
  6 months | 3.30 (1.09) | 3.23 (1.29)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 3.36 (1.11) | 3.39 (1.31)

20. Secondary Outcome: Controlled Motivation as Assessed by the Treatment Self-Regulation Questionnaire for Exercise
Description: as for outcome 19
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
score on a scale
  baseline: number analyzed (Participants) | 152 | 159
  baseline | 3.20 (1.23) | 3.06 (1.25)
  6 months: number analyzed (Participants) | 100 | 104
  6 months | 3.28 (1.24) | 3.29 (1.31)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 3.17 (1.16) | 3.28 (1.27)

21. Secondary Outcome: Amotivation as Assessed by the Treatment Self-Regulation Questionnaire for Diet
Description: Amotivation measured at baseline, 6 months, and 12 months as assessed by the Treatment Self-Regulation Questionnaire (self-administration). This is a 15-item survey scored on a 7 point likert scale from 1 (not at all true) to 7 (very true). Mean score between 1 and 7 will be reported with higher scores indicative of increased amotivation.
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
score on a scale
  baseline: number analyzed (Participants) | 152 | 159
  baseline | 2.30 (1.11) | 2.37 (1.09)
  6 months: number analyzed (Participants) | 100 | 104
  6 months | 2.29 (1.04) | 2.45 (1.16)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 2.47 (1.12) | 2.35 (1.09)

22. Secondary Outcome: Amotivation as Assessed by the Treatment Self-Regulation Questionnaire for Exercise
Description: as for outcome 21
Time Frame: baseline, 6 month, and 12 month follow-up
Population: participants lost to follow up, withdrew, and/or removed from study per physician
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Clinical Care
Number analyzed (Participants) | 157 | 159
score on a scale
  baseline: number analyzed (Participants) | 152 | 159
  baseline | 2.27 (1.09) | 2.31 (1.08)
  6 months: number analyzed (Participants) | 100 | 104
  6 months | 2.27 (1.07) | 2.46 (1.18)
  12 months: number analyzed (Participants) | 86 | 90
  12 months | 2.55 (1.17) | 2.34 (1.08)

23. Other Pre Specified Outcome: Health Coach Fidelity to the Study Intervention
Description: Evaluation of health coach fidelity to administering the motivational interviewing intervention per protocol will be assessed every 2 months using a modified Behavior Change Counseling Index
Time Frame: through completion of administering the study intervention, an average of 4 years
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Adverse Events
Description: Number and type of adverse events
Time Frame: Through study completion, an average of 5 years
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Serious Adverse Events
Description: Number and type of serious adverse events
Time Frame: Through study completion, an average of 5 years
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Withdrawal
Description: Subject Withdrawal Rate
Time Frame: Through study completion, an average of 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 13 months
Description: Participants were asked about Adverse Events (AE) during all in-person visits and by phone in the follow-up call. Participants in the intervention arm were asked about ER, urgent care, hospitalizations, and blood pressure-related symptoms during health coach calls.
Arm/Group | Intervention | Usual Clinical Care
All-Cause Mortality (participants affected / at risk) | 0/157 | 1/159
Serious Adverse Events (participants affected / at risk) | 3/157 | 5/159
Other Adverse Events (participants affected / at risk) | 56/157 | 38/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=157) | Usual Clinical Care (N=159)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 1 (1)
(Gastrointestinal disorders) | 1 (1) | 0 (0)
(Infections and infestations) | 2 (3) | 0 (0)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vascular disorders - Other (Vascular disorders) | 0 (0) | 1 (1)
(General disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=157) | Usual Clinical Care (N=159)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 2 (2)
(Ear and labyrinth disorders) | 1 (1) | 2 (2)
Endocrine disorders - Other (Endocrine disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3 (4) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0)
Immune system disorders - Other (Immune system disorders) | 1 (4) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 5 (7) | 4 (5)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (7)
Nervous system disorders - Other (Nervous system disorders) | 4 (5) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 26 (29) | 15 (19)
Social circumstances - Other (Social circumstances) | 0 (0) | 1 (1)
(Surgical and medical procedures) | 1 (1) | 0 (0)
Vascular disorders - Other (Vascular disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) | 0 (0)
(Cardiac disorders) | 1 (1) | 0 (0)
(Gastrointestinal disorders) | 2 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 2 (2) | 2 (2)
(General disorders) | 1 (1) | 2 (2)
(Infections and infestations) | 6 (9) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (2) | 0 (0)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
(Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
(Metabolism and nutrition disorders) | 1 (1) | 0 (0)
(Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
(Nervous system disorders) | 2 (3) | 0 (0)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
(Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
(Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT03158051/Prot_SAP_000.pdf